CLINICAL TRIAL: NCT02651363
Title: Incidence of Adverse Events, Risk Factors, and Drug Utilization Factors Related to Treatment With Diclofenac 25 MG/Paracetamol 500 MG and Diclofenac 50 MG/Paracetamol 500 MG in Patients From Metropolitan Lima
Brief Title: Diclofenac 25mg/Paracetamol 500 mg and Diclofenac 50 mg/Paracetamol 500 mg for Patients With Pain
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CN003-001
Record Dates: First submitted 2015-12-10; First posted 2016-01-11 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with Dolocordralan

SUMMARY:
The purpose of this study is to collect adverse events and identify risk factors in patients that are taking Dolocordralan Extra 25® and Dolocordralan Extra Forte®

ELIGIBILITY:
Inclusion Criteria:

* Patients who are prescribed Dolocordralan Extra 25 and Dolocordralan Extra Forte at any of the participating clinics
* Patients who sign the informed consent form
* Patients who agree to comply with the study procedures

Exclusion Criteria:

* Please see the protocol for further information on exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or and older from 6 medical centers from Metropolitan Lima, Peru who received at least one dose of Dolocordralan Extra 25 or Dolocordralan Extra Forte according to product label indications will be included in this study
Sampling Method: Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence rate of adverse events (AEs) in patients receiving treatment with Dolocordralan Extra 25 and and Dolocordralan Extra Forte in patients from Metropolitan Lima records | Approximately 13 months
  Ongoing events will be followed up until event resolution

SECONDARY OUTCOMES:
Observed AEs in patients receiving treatment with Dolocordralan Extra 25 and Dolocordralan Extra Forte in patients from Metropolitan Lima records | Approximately 13 months
Risk factors in patients experiencing adverse events while receiving treatment with Dolocordralan Extra 25 and Dolocordralan Extra Forte in patients from Metropolitan Lima records | Approximately 13 months
  Risk factors: medical history, concomitant diseases and concomitant treatment
Drug utilization factors in patients receiving treatment with Dolocordralan Extra 25 and Dolocordralan Extra Forte in patients from Metropolitan Lima records | Approximately 13 months
  Drug utilization factors: Dosing frequency, intake conditions, storage, and concomitant medications

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, San Miguel, Lima region, Peru

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx